CLINICAL TRIAL: NCT05948267
Title: The Effect of Ketamine - Dexmedetomidine Admixture (Ketodex) on Hemodynamic Stability During Anesthesia Induction in Adults: A Randomized Controlled Comparison of Two Doses
Brief Title: The Effect of Ketamine - Dexmedetomidine Admixture (Ketodex) on Hemodynamic Stability During Anesthesia Induction in Adults.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Amany Ahmed Eissa, lecturer of anesthesia& ICU, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MS-94-2023
Record Dates: First submitted 2023-06-15; First posted 2023-07-17 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: The Effect of Ketamine - Dexmedetomidine Admixture (Ketodex) on Hemodynamic Stability
Keywords: ketamine-dexmeditomedine mixture; ketodex; general anesthesia; hemodynamic stability; anesthesia induction
MeSH Terms: interventions — Propofol; Lidocaine; Fentanyl

STUDY DESIGN:
Intervention Model Description: The patients will be divided into 3 equal groups: Propofol group (p), Ketamine-Dexmedetomidine (KD5) group and Ketamine-Dexmedetomidine (KD3) group.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Propofol (P) group (Active Comparator): Propofol(2mg/kg) prepared as will be mixed with 2 mL Lidocaine (40 mg) for concentration 10mg/ml and fentanyl (1mic/kg) prepared for concentration 10mg/ml in 2 separate syringes.
  Interventions: Drug: Propofol, Lidocaine and fentanyl
- Ketamine-Dexmedetomidine (KD5) group (Active Comparator): ketamine (1mg/kg) prepared for concentration 10mg/ml, Dexmedetomidine (0.5microg/kg slow IV) prepared for concentration of 5mic /ml in 2 separate syringes.
  Interventions: Drug: ketamine- dexmeditomidine admixure
- Ketamine-Dexmedetomidine (KD3) group (Active Comparator): ketamine (1mg/kg) prepared concentration 10mg/ml, Dexmedetomidine (0.3microg/kg slow IV) prepared for concentration of 3mic /ml in 2 separate syringes.
  Interventions: Drug: ketamine- dexmeditomidine admixure

INTERVENTIONS:
Drug: ketamine- dexmeditomidine admixure — ketamine in anesthetic dose mixed with two different doses of dexmeditomidine
  Arms: Ketamine-Dexmedetomidine (KD3) group; Ketamine-Dexmedetomidine (KD5) group
Drug: Propofol, Lidocaine and fentanyl — Propofol (2mg/kg) prepared as will be mixed with 2 mL Lidocaine (40 mg) for concentration 10mg/ml and fentanyl (1mic/kg) prepared for concentration 10mg/ml
  Arms: Propofol (P) group

SUMMARY:
The aim of our study to compare two different doses of Dexmedetomidine added to anesthetic dose of ketamine in the induction of general anesthesia in adult patients regarding the hemodynamic profile, adequacy of hypnosis, intubation conditions and recovery type.

We hypothesize that the use of Ketodex during induction of general anesthesia will produce better control regarding the hemodynamic profiles and quality of intubation than propofol.

DETAILED DESCRIPTION:
A randomized, double-blinded, controlled trial. All adult patients (ASA I and II), aged > 18 years old undergoing elective general surgery and meeting the inclusion criteria will be included in the study.

The patients will be divided into 3 equal groups: Propofol group (p), Ketamine-Dexmedetomidine (KD5) group and Ketamine-Dexmedetomidine (KD3) group.

In the operating room; Baseline preoperative arterial pressures (systolic, mean& diastolic) will be the mean of 3 consecutive readings with 30 seconds apart, recorded in the supine position. HR and oxygen saturation baseline will also be recorded.

drug preparation: Propofol (P) group: Propofol(2mg/kg) prepared as will be mixed with 2 mL Lidocaine (40 mg) for concentration 10mg/ml and fentanyl (1mic/kg) prepared for concentration 10mg/ml in 2 separate syringes.

Ketamine-Dexmedetomidine (KD5) group: ketamine (1mg/kg) prepared for concentration 10mg/ml, Dexmedetomidine (0.5microg/kg slow IV) prepared for concentration of 5mic /ml in 2 separate syringes.

Ketamine-Dexmedetomidine (KD3) group: ketamine (1mg/kg) prepared concentration 10mg/ml, Dexmedetomidine (0.3microg/kg slow IV) prepared for concentration of 3mic /ml in 2 separate syringes.

induction of anesthesia: After 3-minutes of preoxygenation, the patients in each group will receive a dose of 0.1ml/Kg boluses of the drugs preparations until achieving clinical loss of consciousness (defined as no response to auditory command and the disappearance of a patient's eyelash reflex).

After loss of consciousness, atracurium 0.5 mg/kg will be administered over 5 seconds, and tracheal intubation will be done after 3 minutes of ventilation through direct laryngoscopy.

The intubation conditions will be graded by the same anesthetist who performed intubation as excellent, good, or poor.

When the trachea is intubated, mechanical ventilation will be applied to obtain SpO2 > 95% and end-tidal CO2 between 30-40 mmHg, and anesthesia will be maintained by 1% isoflurane in air/oxygen admixture. Atracurium maintenance dose of 10 mg will be administered every 20 minutes for maintenance of muscle relaxation.

Any incidence of hypotension (defined as MBP <65 mmHg) will be recorded 20 min after induction. Any episode of hypotension (mean arterial <65 mmHg) will be managed by incremental doses of intravenous ephedrine 5 mg (which will be repeated if hypotension persists for 2 minutes).

Hypertension and tachycardia are defined as mean arterial pressure or heart rate >20% of baseline, respectively. Persistent hypertension (blood pressure increasing after one measurement) will be managed by intravenous 0.25 mg/kg propofol in all groups. Bradycardia (heart rate < 50 bpm) will be managed by 0.5 mg of intravenous atropine.

d. post-operative : After recovery of the patient we will record the Incidence of emergence agitation, Recovery time, the modified Alderet score system for postoperative recovery and the incidence of Postoperative Complications (nausea &vomiting).

The total modified Aldrete score values range from 0 to 12. Scores closer to 0 indicate that the patient is closest to the anesthesia state , Scores of 9 and above indicate that the patient can be discharged and the closer the score is to 12, the higher the chances for all anesthetic, regardless of administering method, to have worn off.

Study outcomes:

1. Primary outcome:

   Incidence of post-induction hypotension defined as a mean arterial pressure MAP < 65 mmHg and/or≤ 70% of baseline reading for > 10 s within the first 20 min after general anesthesia induction.
2. Secondary outcome:

Mean arterial pressure, SBP, DBP, heart rate at baseline, immediately after induction, after intubation, then every 2-minute till skin incision.

Total Ephedrine requirements during the period from induction anesthesia to skin incision.

Total Atropine requirements during the period from induction anesthesia to skin incision.

Severe post-induction hypotension (mean arterial pressure ≤60 mmHg), hypertension, bradycardia, and tachycardia during 30 min from induction anesthesia.

The Number of hypotensive episodes. Intubation time (time from insertion of the laryngoscope into the mouth until its removal after tracheal intubation) Response to intubation score. Total dexmedetomidine, ketamine and propofol dose per weight. Recovery time Incidence of emergence agitation using Riker Sedation-Agitation Scale

Statistical analysis:

Sample size justification The incidence of post induction hypotension in a previous study (10) for the control group was 58%. At alpha error of 0.05, we calculated that 96 patients would give 80% power to detect 30% absolute reduction in the incidence of hypotension in the treatment group. However, to allow the comparisons between the control group and each treatment group, an adjusted P (Bonferroni correction) of 0.025 was set for the primary outcome and the required sample size increased to 114 patients (38 patients per group). The number of prepared envelopes will be 123 (41 envelopes per group) to compensate for possible dropouts. The sample size was calculated using MedCalc Software version 14 (MedCalc Software bvba, Ostend, Belgium).

Statistical methods The collected data will be coded, tabulated, and statistically analyzed using IBM SPSS statistics (Statistical Package for Social Sciences) software version 22.0, IBM Corp., Chicago, USA, 2013. Quantitative data will be described as mean±SD (standard deviation) and then compared using an independent t-test. Qualitative data will be described as numbers and percentages and compared using the Chi-square test. The level of significance will be taken at p-value < 0.050 is significant, otherwise is non-significant.

ELIGIBILITY:
Inclusion Criteria:

- All patients undergoing elective general surgery. Patients aged >18 years. ASA I and II. Both sexes.

Exclusion Criteria:

* All patients undergoing emergency surgery. Patients less than 18 years. History of difficult intubation, abnormal airway examination Cardiac morbidities (impaired contractility with ejection fraction < 50%, heart block, arrhythmias, tight valvular lesions).

Patients on angiotensin converting enzyme inhibitors and angiotensin receptor blockers medications.

Patients with uncontrolled hypertension. Patients with allergy of any of the study drugs. Body mass index > 35 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Incidence of post-induction hypotension | the first 20 min after general anaesthesia induction.
  mean arterial pressure MAP < 65 mmHg and/or≤ 70% of baseline reading for > 10 s

SECONDARY OUTCOMES:
Total Ephedrine requirements | during the period from induction anesthesia to skin incision. maximum 30 minutes
Total Atropine requirements | during the period from induction anesthesia to skin incision. max 30 minutes
Severe post-induction hypotension (mean arterial pressure ≤60 mmHg), hypertension, bradycardia, and tachycardia | during 30 min from induction anesthesia.
The Number of hypotensive episodes | the 2 hours procedure
Intubation time (time from insertion of the laryngoscope into the mouth until its removal after tracheal intubation) | maximum 5 minutes
  (time from insertion of the laryngoscope into the mouth until its removal after tracheal intubation) (time from insertion of the laryngoscope into the mouth until its removal after tracheal intubation)
Response to intubation score. | maximum 5 minutes
Total dexmedetomidine, ketamine and propofol dose per weight. | the whole procedure . 2 hours
Recovery time | less than 15 minutes
Incidence of emergence agitation using Riker Sedation-Agitation Scale | 60 minutes

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Kasr Al Ainy Hospitals, Cairo
  - Kasr Alainy Hospitals Cairouniversity, Cairo

IPD SHARING:
Plan to Share IPD: No